CLINICAL TRIAL: NCT05373121
Title: Is Signposting to Online Peer Support Helpful in Decreasing Loneliness in Parents of Children With Long-term Conditions and Disabilities? A Randomised Controlled Trial
Brief Title: Is Signposting to Online Peer Support Helpful in Decreasing Loneliness in Parents of Children With Long-term Conditions and Disabilities?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22125/001
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Loneliness; Anxiety; Anxiety Disorder; Depression; Low Mood
Keywords: randomised controlled trial; loneliness; peer support; online peer support; long-term condition; chronic illness; parenting
MeSH Terms: conditions — Anxiety Disorders; Depression; Consciousness Disorders; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention condition - signposting to online peer support (Experimental): The intervention group will be sent a list of online peer support signposting groups and forums to engage with, which will be adapted depending on what health conditions their child has. They will be asked to keep a weekly engagement log for three months.
  Interventions: Behavioral: Online Peer Support
- Waitlist condition (No Intervention): The waitlist group will be informed that they will be contacted again in three months, after which, the waitlist will be sent the signposting resources.

INTERVENTIONS:
Behavioral: Online Peer Support — Signposting to online peer support groups and forums
  Arms: Intervention condition - signposting to online peer support

SUMMARY:
The present study aims to evaluate whether signposting to online peer support will be associated with a significant decrease in self-reported loneliness for parents of children with long-term conditions and disabilities. Parents of children with long-term conditions and disabilities will be randomised to either the treatment condition, being signposted to online peer support, or to the waitlist condition. Whether signposting to online peer support has an impact on social capital and anxiety and depression will also be investigated.

DETAILED DESCRIPTION:
Loneliness has been defined as an aversive subjective experience that occurs when a person's social network is lacking in either quality or quantity compared to their needs. A recent poll of 2000 parents found that more than half had experienced a problem with loneliness.

There is ample evidence that parental loneliness has negative consequences for both the parent and child. Loneliness has been associated with parental stress, with maternal loneliness being associated with dissatisfaction with life and the couple relationship and depressive symptoms, and found to be a predictor of chronic depression. Paternal loneliness has been shown to predict son's loneliness, and daughter's loneliness is predicted by maternal loneliness. Additionally, maternal loneliness has been found to predict social competence and fear of negative evaluation in adolescents.

Social capital, which has been defined as the creation of personal relationships and the benefits that come with them, has been found to be significantly inversely associated with loneliness in different populations, for example older adults and students.

A recent scoping review found that parents of children with long-term conditions or disabilities appear to be at increased risk of loneliness, but there has been little research looking directly at what might help to alleviate loneliness in this group. The review identified that peer support could be a potential key mechanism in reducing loneliness in parents.

With stretched mental health services for families in the UK, parents are often signposted to peer support groups for advice and support. Due to the COVID-19 pandemic many face-to-face peer support groups have been forced to close, with signposting options being limited to online peer support groups or forums.

The primary aim of the study is to evaluate the effectiveness of signposting parents of children with long-term conditions and disabilities to peer support groups in terms of alleviating loneliness (relative to a wait list control). A secondary aim is to identify the predictors of such change / any response to allocation to the peer support groups, including attendance of the peer support and changes in online and offline social capital. Whether signposting to online peer support has an impact on anxiety and depression will also be investigated.

ELIGIBILITY:
Inclusion criteria:

* participants will be required to have one or more child with long-term conditions or disabilities
* participants must consent to take part
* participants should be sufficiently fluent in English to enable participation in online peer support groups and forums as well as participation in the study.

Exclusion criteria:

- participants must not be under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Loneliness | Measured at baseline (time 1), post (3 months - time 2), follow up (6 months - time 3)
  Change in self-reported loneliness on the 20-item revised UCLA Loneliness Scale (R-UCLA: Russell, Peplau, & Cutrona, 1980). Scores range from 20 to 80, with higher scores indicating a higher level of self-reported loneliness.

SECONDARY OUTCOMES:
Social Capital | Measured at baseline (time 1), post (3 months - time 2), follow up (6 months - time 3)
  Change in self-reported social capital (online and offline) on the Williams' (2006) Internet Social Capital scale. Scores range from 10 to 50 on each subscale (online and offline), with higher scores indicating a higher level of self-reported social capital
Anxiety and Depression | Measured at baseline (time 1), post (3 months - time 2), follow up (6 months - time 3)
  Change in self-reported anxiety and depression on the Hospital Anxiety and Depression Scale (Zigmond & Snaith, 1983). Scores range from 0-21 on each subscale (depression and anxiety), with higher scores indicating a higher level of self-reported anxiety or depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Bennett, Principal Investigator — University College, London
Locations (1):
- University College, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be stored indefinitely on a secure UCL database and may be used for future research, it will not be identifiable to you in any way.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: Data will be available on reasonable request

REFERENCES:
- [Background] Au A, Chan YC, Cheung G, Yuen P, Lee T. Examining the correlation between parenting stress and social support and loneliness in Chinese mothers living in a socially impoverished community in Hong Kong. Journal of Psychology in Chinese Societies. 2008 Jul 1;9(2):167.
- [Background] Action for Children. It starts with hello: A report into the impact of loneliness in children, young people and families. London; 2017
- [Background] Bai Z, Wang Z, Shao T, Qin X, Hu Z. Association between social capital and loneliness among older adults: a cross-sectional study in Anhui Province, China. BMC Geriatr. 2021 Jan 7;21(1):26. doi: 10.1186/s12877-020-01973-2. PMID 33413141
- [Background] Perlman D, Peplau LA. Loneliness research: A survey of empirical findings. Preventing the harmful consequences of severe and persistent loneliness. 1984;13:46.
- [Background] Luoma I, Korhonen M, Puura K, Salmelin RK. Maternal loneliness: concurrent and longitudinal associations with depressive symptoms and child adjustment. Psychol Health Med. 2019 Jul;24(6):667-679. doi: 10.1080/13548506.2018.1554251. Epub 2018 Dec 5. PMID 30514104
- [Background] Luoma I, Korhonen M, Salmelin RK, Helminen M, Tamminen T. Long-term trajectories of maternal depressive symptoms and their antenatal predictors. J Affect Disord. 2015 Jan 1;170:30-8. doi: 10.1016/j.jad.2014.08.017. Epub 2014 Aug 30. PMID 25218734
- [Background] Salo AE, Junttila N, Vauras M. Social and emotional loneliness: Longitudinal stability, interdependence, and intergenerational transmission among boys and girls. Family Relations. 2020 Feb;69(1):151-65.
- [Background] Zafar N, Kausar R. Psychosocial implications of early father separation for adolescents and their mothers. Age. 2015;47(5).
- [Background] Williams D. On and off the'Net: Scales for social capital in an online era. Journal of computer-mediated communication. 2006 Jan 1;11(2):593-628.
- [Background] Nowland R, Thomson G, McNally L, Smith T, Whittaker K. Experiencing loneliness in parenthood: a scoping review. Perspect Public Health. 2021 Jul;141(4):214-225. doi: 10.1177/17579139211018243. PMID 34286652